CLINICAL TRIAL: NCT02683668
Title: Targeting of the Small Airways in Patients With COPD: Airway Effects of Tiotropium - Respimat vs Handihaler
Brief Title: Airway Effects of Tiotropium in Patients With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 151C2697
Record Dates: First submitted 2016-02-11; First posted 2016-02-17 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: COPD; LUNG DISEASES, OBSTRUCTIVE
Keywords: Inhalers; Tiotropium
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive

STUDY DESIGN:
Intervention Model Description: Each volunteer get all treatment in a same sequence
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Handihaler-Tiotropium 18 mcg untrained (Experimental): Patients receiving Handihaler who have not been trained (real-life use) for over 3 months on its use. Here the investigators want to see that if patients have on-going symptoms but are on Handihaler-Tiotropium 18mcg what is happening PRIOR to proper inhaler technique training - that is their 'real-life' use of the inhaler - to their lung function (large and small airways) and also symptoms or exercise limitation (determined by CAT score) will already be recorded as entry criteria
  Interventions: Combination Product: Handihaler-Tiotropium 18 mcg untrained
- Handihaler-Tiotropium 18 mcg trained (Experimental): Patients will be trained in their use of Handihaler-Tiotropium and asked to take 18 mcg once daily for 14 days to see if their (i) airway lung function and or (ii) clinical symptoms improve. Here the investigators want to see what happens AFTER proper inhaler technique training on large and small airways lung function and also symptoms or exercise limitation (determined by CAT score)
  Interventions: Combination Product: Handihaler-Tiotropium 18 mcg trained
- Respimat-Tiotropium 5 mcg trained (Experimental): Patients will be switched to trained Respimat Tiotropium 5 mcg once daily for 14 days to see if their (i) airway lung function and or (ii) clinical symptoms improve. Here the investigators want to see what happens AFTER this efficient device Respimat (trained) compared to PREVIOUS device Handihaler (trained) on large and small airways lung function and also symptoms or exercise limitation (determined by CAT score). The investigators want to see if the properties of the Respimat device with deeper lung deposition (slow velocity and small particles) can improve small airway measures (and indeed large airway measures) that might also be related to an improvement in symptoms.
  Interventions: Combination Product: Respimat-Tiotropium 5 mcg trained

INTERVENTIONS:
Combination Product: Handihaler-Tiotropium 18 mcg untrained — We are looking at the untrained used of Handihaler
  Arms: Handihaler-Tiotropium 18 mcg untrained
Combination Product: Handihaler-Tiotropium 18 mcg trained — We are looking at the trained use of Handihaler after 14 days treatment
  Arms: Handihaler-Tiotropium 18 mcg trained
Combination Product: Respimat-Tiotropium 5 mcg trained — we are looking at the trained use of Respimat after 14 days treatment
  Arms: Respimat-Tiotropium 5 mcg trained

SUMMARY:
The aim of the study is to investigate the effect of tiotropium from different devices on a panel of small (IOS, MBNW, DLCO, FVC) and large airway (FEV1, PEF) responses in patients with mild-moderate COPD. Comparisons will be made between Tiotropium Handihaler 18 micrograms once daily and Tiotropium Respimat 5 micrograms once daily

DETAILED DESCRIPTION:
Patients with asthma and chronic obstructive airways disease (COPD) undergo routine testing of their lung function in the diagnosis, progression, management and, response to treatment of their disease. Standard lung function obtains measurements based on the forced flow of air moving within the airways. Such measurements give a reasonable assessment of disease affecting the large airways, but not an accurate estimate of small airways disease. Small airways are less than 2mm in diameter. However, both asthma and COPD have disease that involves not only the large but also the small airways that has important clinical consequences. Indeed, COPD predominantly affects the small airways.

Tiotropium (Spiriva, Boehringer Ingelheim), a long-acting inhaled anticholinergic bronchodilator, improves lung function, quality of life, and exercise endurance and reduces exacerbations in patients with chronic obstructive pulmonary disease (COPD).

Respimat Soft MistTM Inhaler (SMI) is a novel inhaler delivering a unique slow-moving Soft MistTM that allows gentle inhalation - making it easy to inhale. Importantly it has drug particles that are ~ 2microns that allow an increase in the total lung deposition of drug (~52%) and also the potential for penetration to treat the small and large airways in patients with COPD; that is targeting the whole airway tree.

RESEARCH AIM & HYPOTHESIS The aim is to investigate the effect of tiotropium from different devices on a panel of small (IOS, MBNW, DLCO, FVC) and large airway (FEV1, PEF) responses in patients with mild-moderate COPD. The investigators will compare Tiotropium Handihaler 18 micrograms once daily with Tiotropium Respimat 5 micrograms once daily.

The investigators will identify a COPD cohort with ongoing symptoms or exercise limitation on HandiHaler, as proposed. The science behind this is why are people still limited (even if partially as determined using the CAT score) and is more distal airway targeting necessary? This doesn't necessarily mean targeting the acinar/alveolar beyond the terminal bronchioles, but just a little bit deeper into the distal conducting airway. This can be achieved with Respimat.

ELIGIBILITY:
Inclusion Criteria:

1. COPD patients with FEV1/FVC <70% predicted.
2. Mild (GOLD stage I: FEV1 >80% pred.) to moderate (GOLD stage II: FEV1 50-80% pred.)
3. Aged 30 years onwards - there is no upper age limit as we do not want to exclude elderly patients as COPD is primarily a disease in the elderly population.
4. Have on-going symptoms or exercise limitation (determined by CAT score)
5. Stable COPD (no chest infection requiring antibiotics and/or oral steroids in the past 2 months).
6. Capable of giving informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

1. Subjects who lack the capacity to consent will not be recruited.
2. Current or past diagnosis of asthma.
3. Patients on concurrent oral bronchodilators (theophylline, PDE4 inhibitors) will not be included.
4. Patients on other LAMAs will not be included
5. History of any chronic respiratory diseases other than COPD.
6. History of another medical condition, which in the opinion of the Unit Physician, contraindicates his/her participation in the study.
7. Clinical evidence of heart failure (NYHA class III-IV).
8. Unstable respiratory disease in the last four weeks prior to the screening visit (indicated by any change in their maintenance inhaled therapy or who have had a lower respiratory tract infection in the previous four weeks).
9. Evidence of a respiratory exacerbation requiring emergency room treatment and/or hospitalisation within four weeks before screening.
10. Use of systemic (oral or intravenous) steroids 4 weeks prior to inclusion (injectable depot steroids 6 weeks) or more than 3 periods during the last 12 months.
11. Participants with a known or suspected allergy, sensitivity or intolerance to the study drugs (this will be asked directly at the screening visit) or patients with a history of another drug allergy which, in the opinion of the Unit Physician, contraindicates his/her participation in the study.
12. Patients with known or suspected cardiac rhythm disorders
13. Patients treated with beta-blockers in the week preceding the screening visit and during the study period.
14. Females who are pregnant or lactating or are likely to become pregnant during the trial. (a urine pregnancy test will be performed. Women of childbearing potential may be included in the study if, in the opinion of the investigator, they are taking adequate contraceptive precautions.
15. Patients who have evidence of alcohol or substance abuse.
16. Participation in another clinical trial with an investigational drug in the four weeks preceding the screening visit.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omar Usmani, Principal Investigator — Imperial College London
Locations (1):
- Asthma Lab, Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-four subjects (23 male) with mild-to-moderate COPD (GOLD stage I-II, FEV1 67.8% of predicted) using DPI-HandiHaler (18µg tiotropium daily) for at least 3 months, but with ongoing symptoms or exercise limitation (COPD Assesment Test (CAT) score >10) participated in the study. 1 failed to complete
Period: Period 1
Arm/Group | Handihaler-Tiotropium 18 mcg Untrained | Handihaler-Tiotropium 18 mcg Trained | Respimat-Tiotropium 5 mcg Trained
Started | 44 | 0 | 0
Completed | 44 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Period 2
Arm/Group | Handihaler-Tiotropium 18 mcg Untrained | Handihaler-Tiotropium 18 mcg Trained | Respimat-Tiotropium 5 mcg Trained
Started | 0 | 44 | 0
Completed | 0 | 43 | 0
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Period: Period 3
Arm/Group | Handihaler-Tiotropium 18 mcg Untrained | Handihaler-Tiotropium 18 mcg Trained | Respimat-Tiotropium 5 mcg Trained
Started | 0 | 0 | 43
Completed | 0 | 0 | 43
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participant: Patients receiving Handihaler who have not been trained (real-life use) for over 3 months on its use.
Arm/Group | All Participant
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 44
R5 - R20 (Peripheral Airways Resistance) [Mean (Standard Deviation); unit: kPa/l/s] | 0.608 (0.207)

OUTCOME MEASURES:

1. Primary Outcome: Peripheral Airways Resistance (R5-R20)
Description: Peripheral airways resistance measured by impulse oscillometry (IOS). Specific frequencies relate to different levels: a frequency of 5 hertz (Hz) provides values for total airway resistance (R5) and reactance (X5); a 20Hz frequency gives a value for central or large airway resistance (R20); and if one subtracts the value of central airway resistance from that for total airway resistance (i.e. R5-R20), this provides a measure of peripheral or small airways resistance.
Time Frame: 28 days
Measure: Mean (Full Range); unit: kPa/l/s
Arm/Group | Handihaler-Tiotropium 18 mcg Untrained | Handihaler-Tiotropium 18 mcg Trained | Respimat-Tiotropium 5 mcg Trained
Number analyzed (Participants) | 44 | 43 | 43
kPa/l/s | 0.23 [0.004 to 0.56] | 0.2 [0.03 to 0.62] | 0.16 [0.03 to 0.42]

2. Secondary Outcome: Sacin
Description: Multiple Breath Nitrogen Washout (MBNW). Sacin is a gas exchange measures, assessing convectional ventilation heterogeneity in pre acinar/acinar airways.
Time Frame: 28 days
Measure: Mean (Full Range); unit: kPa\l\s
Arm/Group | Handihaler-Tiotropium 18 mcg Untrained | Handihaler-Tiotropium 18 mcg Trained | Respimat-Tiotropium 5 mcg Trained
Number analyzed (Participants) | 44 | 43 | 43
kPa\l\s | 0.333 [0.11 to 0.53] | 0.339 [0.06 to 0.57] | 0.345 [0.03 to 0.65]

3. Secondary Outcome: Lung Function FEV1
Description: Lung function parameters FEV1
Time Frame: 28 days
Measure: Mean (Full Range); unit: liters
Arm/Group | Handihaler-Tiotropium 18 mcg Untrained | Handihaler-Tiotropium 18 mcg Trained | Respimat-Tiotropium 5 mcg Trained
Number analyzed (Participants) | 44 | 43 | 43
liters | 1.575 [0.72 to 2.67] | 1.58 [0.51 to 2.56] | 1.651 [0.74 to 2.65]

4. Secondary Outcome: Scond
Description: MBW parameters. Scond is a gas exchange measures, assessing convectional ventilation heterogeneity in peripheral conducting airways.
Time Frame: 28 days
Measure: Mean (Full Range); unit: kPa\l\s
Arm/Group | Handihaler-Tiotropium 18 mcg Untrained | Handihaler-Tiotropium 18 mcg Trained | Respimat-Tiotropium 5 mcg Trained
Number analyzed (Participants) | 44 | 43 | 43
kPa\l\s | 0.05 [0.011 to 0.17] | 0.04 [0.01 to 0.12] | 0.04 [0 to 0.12]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | All Participant
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-09-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT02683668/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT02683668/SAP_001.pdf